CLINICAL TRIAL: NCT07264205
Title: Safety and Feasibility Study of RT-310 for Treatment of Lower Urinary Tract Symptoms (LUTS) Secondary to Benign Prostatic Hyperplasia (BPH)
Brief Title: RT-310 Safety and Feasibility BPH Study
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Resurge Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P18003
Record Dates: First submitted 2025-11-24; First posted 2025-12-04 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-11

CONDITIONS: BPH (Benign Prostatic Hyperplasia)
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- RT-310 (Experimental): RT-310
  Interventions: Combination Product: RT-310

INTERVENTIONS:
Combination Product: RT-310 — RT-310

SUMMARY:
RT-310, is intended to deliver drug locally to the prostate gland for the management of prostate disease, while minimizing systemic exposure and its associated side-effects. The objectives of the study are to assess whether RT-310 is safe and feasible for the participant population.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Diagnosis of symptomatic BPH
* Age ≥ 50 years up to 80 years
* International Prostate Symptom Score (IPSS) ≥ 13
* Peak urine flow rate ≥ 5mL/sec and ≤ 12 ml/sec, voided volume ≥ 100 ml
* Prostate volume 30 to 80 cc per ultrasound
* Post void residual (PVR) urine ≤ 250 ml
* Inadequate response and/or refusal of medical therapy for LUTS

Exclusion Criteria:

* Unable or unwilling to sign the informed consent form (ICF) and/or comply with the study follow-up requirements
* Current urinary retention requiring catheterization
* Unwilling to abstain from unprotected sexual intercourse for 3 months
* Unwilling to abstain from any child conceiving activities for 6 months
* Have an obstructive or protruding median lobe of the prostate
* High bladder neck determined by Investigator
* Active urinary tract infection at time of treatment
* Previous BPH surgical procedure or implants, urethral stricture, Any prior minimally invasive intervention (e.g. TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
* Previous pelvic surgery or irradiation
* History of neurogenic or atonic bladder
* Stress urinary incontinence, mixed or urge incontinence
* Biopsy of the prostate within the past 6 weeks
* Life expectancy estimated to be less than 1 year
* History of prostate or bladder cancer, confirmed or suspected malignancy of prostate or bladder
* History of compromised renal function or upper urinary tract disease
* Known coagulopathies or participant on anticoagulants or antiplatelets other than aspirin ≤ 100 mg (unless antiplatelets are withheld minimum 3 days prior to procedure)
* Use of the following medications pre-screening:

Within 6 months of baseline assessment, unless documented on stable dose for ≥ 12 months: 5-alpha-reductase inhibitors (e.g. dutasteride, Avodart, finasteride, Proscar, Propecia) Within 4 months of baseline assessment: estrogen, any drug producing androgen suppression, or anabolic steroids Within 2 weeks of baseline assessment: alpha-blockers, gonadotropin- releasing hormonal analogs, anticholinergics or cholinergic medication or phenylephrine, pseudoephedrine, diphenhydramine or imipramine medications Within 1 week of baseline assessment, unless documented on stable dose for ≥ 6 months: beta blockers, antidepressants, anticonvulsants, and antispasmodics

* Cystolithiasis within the prior 3 months
* History of co-morbidities that would affect having an elective urological procedure including prostatitis, conditions that preclude the RT-310.
* Other co-morbidities that could impact the study results such as:

Severe cardiac arrhythmias uncontrolled by medications or pacemaker Congestive heart failure New York Heart Association (NYHA) III or IV History of uncontrolled diabetes mellitus Significant respiratory disease in which hospitalization may be required

* Known immunosuppression (i.e. AIDS, post-transplant, undergoing chemotherapy)
* Currently enrolled in any other investigational clinical research trial that has not completed the primary endpoint.
* No more than two documented active urinary tract infections (UTI) by culture or bacterial prostatitis within last year documented by culture (UTI is defined as >100,000 colonies per ml urine from midstream clean catch or catheterization specimen)
* Current gross hematuria and/or visible hematuria with participant urine sample without known contributing factor
* Presence of a penile implant or stent(s) in the urethra or prostate
* PSA > 10 ng/ml unless prostate cancer is ruled out by biopsy. If PSA is > 4 ng/ml and ≤ 10 ng/ml, prostate cancer must be ruled out to the satisfaction of the investigator via additional tests including digital rectal exam (DRE) and/or biopsy
* Active or history of epididymitis within the past 3 months
* Sensitivity to RT-310
* Parkinson's disease or other neurologic disease that may impact bladder function such as stroke, TIA, multiple sclerosis
* Active infection including prostatitis

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 20 (Estimated)
Dates: Start 2025-03-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Safety Endpoint | Baseline to Day 180
  Absence of unanticipated adverse events (UAEs) not listed in the protocol or Adverse Events (AEs) that meet the protocol definition of Serious Adverse Events (SAEs)

SECONDARY OUTCOMES:
Change in IPSS | Baseline to Day 180
  International Prostate Symptom Score (IPSS)
Uroflowmetry (Qmax) | Baseline to Day 180
  Peak Urinary Flowrate (Qmax)

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Santo Domingo, Dominican Republic

IPD SHARING:
Plan to Share IPD: No